CLINICAL TRIAL: NCT01467011
Title: An Open-label Study of the Pharmacokinetics of Mycophenolic Acid as Myfortic (Enteric-coated Mycophenolate Sodium) When Used in Combination With Prograf (Tacrolimus) and Corticosteroids in Patients Undergoing de Novo Liver Transplantation
Brief Title: Myfortic, Prograf, and Corticosteroids in de Novo Liver Transplantation
Status: Completed | Type: Observational
Sponsor: R. Mark Ghobrial, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, R. Mark Ghobrial, MD, Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00004722
Record Dates: First submitted 2011-11-01; First posted 2011-11-08 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: End Stage Liver Disease
Keywords: Myfortic; Mycophenolic acid; Prograf; Tacrolimus; Liver transplantation
MeSH Terms: conditions — End Stage Liver Disease | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be retained and frozen for MPA levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cases: de novo liver transplant recipients receiving Enteric-coated Mycophenolate Sodium
  Interventions: Drug: Enteric-coated Mycophenolate Sodium

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate Sodium — 1440mg/day for 6 months posttransplant
  Other Names: mycophenolic acid

SUMMARY:
The purpose of this study is to gather information regarding the use of Myfortic, Prograf, and corticosteroids in new liver transplant recipients. These three medicines help to prevent the body from rejecting the transplanted liver. The information the investigators are obtaining is data relating to the process of Myfortic absorption by the body, its distribution in the body, the breakdown of Myfortic in the body, and its elimination from the body. This absorption, distribution, breakdown, and elimination is called pharmacokinetics.

DETAILED DESCRIPTION:
Myfortic is approved for use in kidney transplant recipients, and has been prescribed by doctors for liver transplant recipients. No study has been reported to date evaluating the pharmacokinetics of Myfortic in new liver transplant recipients who also take Prograf and corticosteroids. During this six month study, a series of blood samples will be obtained after subjects take Myfortic, Prograf, and corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Adults > or equal to age 18 years
* Planned to receive tacrolimus and corticosteroid therapy posttransplant
* Serum creatinine at transplant < or equal to 2.5mg/dL
* UCSF tumor staging < 8cm total
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the baseline visit and are required to practice a reliable method of contraception for the duration of the study and for no fewer than 6 weeks after completing the study.
* Signed informed consent form prior to any research assessment

Exclusion Criteria:

* Induction therapy
* Requiring dialysis at the time of transplant
* Organ transplant other than liver
* Pregnant or nursing females
* Women of childbearing potential not practicing reliable methods of contraception. Reliable methods for contraception include surgical sterilization (hysterectomy, bilateral tubal ligation), double-barrier method (such as condom and diaphragm). To be considered as post-menopausal and not of childbearing potential, female subjects must have experienced 12 consecutive months of amenorrhea.
* Require any medications that interfere with metabolism of Myfortic (other than corticosteroids)
* Have a known hypersensitivity to mycophenolate sodium, mycophenolic acid, mycophenolate mofetil, or any of its excipients
* Participation in a study of investigational drug in the previous 30 days or 5 half-lives of the investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage liver disease who are receiving a liver transplant at The Methodist Hospital in Houston, Texas and who satify the inclusion/exclusion criteria will be considered for the study.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Twelve hour pharmacokinetics at one week, one month, and six months post transplant
  Pharmacokinetic time points will be obtained at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 8, and 12 hours post dose. The exposure (area under the concentration-time curve, AUC μg·h/mL, Cmax ng/mL, and Tmax, hours) of MPA and MPAG will be calculated using non-compartmental analysis.

SECONDARY OUTCOMES:
Safety and tolerability | 1 week, 1 month, 6 months
  MPA exposure will be assessed at one week, 1 month, and 6 months. Kidney function (using MDRD and Cockcroft-Gault) will be compared with PK parameters and graft survival recorded. Adverse events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: R M Ghobrial, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Background] Plank LD, Metzger DJ, McCall JL, Barclay KL, Gane EJ, Streat SJ, Munn SR, Hill GL. Sequential changes in the metabolic response to orthotopic liver transplantation during the first year after surgery. Ann Surg. 2001 Aug;234(2):245-55. doi: 10.1097/00000658-200108000-00015. PMID 11505071
- [Background] de Carvalho L, Parise ER, Samuel D. Factors associated with nutritional status in liver transplant patients who survived the first year after transplantation. J Gastroenterol Hepatol. 2010 Feb;25(2):391-6. doi: 10.1111/j.1440-1746.2009.06033.x. Epub 2009 Nov 19. PMID 19929929
- [Background] Pisupati J, Jain A, Burckart G, Hamad I, Zuckerman S, Fung J, Venkataramanan R. Intraindividual and interindividual variations in the pharmacokinetics of mycophenolic acid in liver transplant patients. J Clin Pharmacol. 2005 Jan;45(1):34-41. doi: 10.1177/0091270004270145. PMID 15601803
- [Background] Jain A, Venkataramanan R, Hamad IS, Zuckerman S, Zhang S, Lever J, Warty VS, Fung JJ. Pharmacokinetics of mycophenolic acid after mycophenolate mofetil administration in liver transplant patients treated with tacrolimus. J Clin Pharmacol. 2001 Mar;41(3):268-76. doi: 10.1177/00912700122010087. PMID 11269567
- [Background] Arns W, Breuer S, Choudhury S, Taccard G, Lee J, Binder V, Roettele J, Schmouder R. Enteric-coated mycophenolate sodium delivers bioequivalent MPA exposure compared with mycophenolate mofetil. Clin Transplant. 2005 Apr;19(2):199-206. doi: 10.1111/j.1399-0012.2004.00318.x. PMID 15740555
- [Background] Perry TW, Christians U, Trotter JF, Bendrick-Peart J. Pharmacokinetics of enteric-coated mycophenolate sodium in stable liver transplant recipients. Clin Transplant. 2007 May-Jun;21(3):413-6. doi: 10.1111/j.1399-0012.2007.00662.x. PMID 17488394
- [Background] Kaczmarek I, Bigdeli AK, Vogeser M, Mueller T, Beiras-Fernandez A, Kaczmarek P, Schmoeckel M, Meiser B, Reichart B, Ueberfuhr P. Defining algorithms for efficient therapeutic drug monitoring of mycophenolate mofetil in heart transplant recipients. Ther Drug Monit. 2008 Aug;30(4):419-27. doi: 10.1097/FTD.0b013e31817d7064. PMID 18641552